CLINICAL TRIAL: NCT05641727
Title: Plyometric Training Versus Strengthening Exercise On Muscle Strength, Selective Motor Control And Quality Of Life In Children With Hemiplegia
Brief Title: Plyometric Training Versus Strengthening Exercise On Children With Hemiplegia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohammed Alzagh, principal investigator, Cairo University
Other Study IDs: plyometrics on hemiplegia
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Children With Hemiplegic cp; Effect of Plyometic Exercises

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the effect of plyometric training versus strengthening exercise on quadriceps and hamstring muscles and quality of life and selective motor control of lower limb of children with hemiplegia.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effect of plyometric training versus strengthening exercise on quadriceps and hamstring muscles and quality of life and selective motor control of lower limb of children with hemiplegia.

Hand-Held dynamometer is used to assess the muscle strength of quadriceps and hamstring Selective control assessment of lower extremity scale is used to assess selective motor control of lower limb.

Peds Ql scale is used to assess quality of life of the children. The methods of assessment are valid and reliable.

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranging from 8 to 10 years.
* They will be on level (1 : 1+) according to Modified Ashworth scale
* They will be on level I according to Gross Motor Functional Classification System
* They can understand and follow instructions.

Exclusion Criteria:

* Child undergoes orthopedic surgery past one year.
* Visual or auditory problems that interfere with rehabilitation programs.
* Botox injection past 6 months.
* Cardiac problems or uncontrolled seizures.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with hemiplegic cp aged from 8 - 10 years.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | three months
  Muscle strength of quadriceps and hamstrings is assessed by Hand-Held dynamometer
Quality of life of children | three months
  Quality of life of children (physical, psychological and social) is assessed by PedsQl scale PedsQl scale scoring from 0-100 scale The higher scores indicate better health related quality of life and lower scores indicate worse health related quality of life
Selective motor control of lower limb | three months
  Selective motor control of lower limb is assessed by selective control assessment of lower extremity scale The scale has 3 grades for each joint (hip, knee, ankle, sub-talar and toes) 0 point : unable
  1. point : impaired
  2. points : normal

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Abdel-Nabie, phd, Study Chair — assisstant professor of pediatric physical therapy; Amira Ibrahim, phd, Study Chair — lecturer
Locations (1):
- Outpatient Clinic of Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No